CLINICAL TRIAL: NCT00003996
Title: A Phase II Trial of Pre-irradiation Chemotherapy With BCNU, Cisplatin and Oral Etoposide Combined With Radiation Therapy in the Treatment of Grade 4 Astrocytoma (Glioblastoma)
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-987252; NCI-2012-02308 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000067206 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-06-17 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Carmustine; Drug Therapy; Cisplatin; Etoposide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chemotherapy + carmustine + etoposide + cisplatin + radiation (Experimental): Patients receive pre-irradiation chemotherapy consisting of carmustine IV over 1 hour on days 1-3 and oral etoposide on days 1-21 and 29-49 immediately followed by cisplatin IV over 1-2 hours on days 1-3 and 29-31. Treatment repeats every 8 weeks for 2 courses. Patients receive concurrent cranial radiotherapy daily over 8 weeks during course 2. Patients then receive carmustine IV over 1-2 hours every 8 weeks for 4 courses. Treatment continues in the absence of disease progression or unacceptable toxicity. Quality of life is assessed before the study, prior to each treatment course, every 4 months for 1 year, every 6 months for 4 years, and then annually for 5 years. Patients are followed every 4 months for 1 year, every 6 months for 4 years, annually for 5 years, and then for survival.
  Interventions: Drug: carmustine; Drug: chemotherapy; Drug: cisplatin; Drug: etoposide; Radiation: radiation therapy

INTERVENTIONS:
Drug: carmustine
Drug: chemotherapy
Drug: cisplatin
Drug: etoposide
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one chemotherapy drug with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus radiation therapy in treating patients who have newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of carmustine, cisplatin, and etoposide administered prior to and during radiotherapy in patients with newly diagnosed high grade glioblastoma multiforme. II. Assess the toxicities of this treatment regimen in this patient population. III. Assess fatigue, depression, and excessive daytime somnolence in terms of incidence, duration, and relation to age, tumor type, tumor site, cancer therapy, and symptoms in this patient population. IV. Evaluate the quality of life of these patients.

OUTLINE: Patients receive pre-irradiation chemotherapy consisting of carmustine IV over 1 hour on days 1-3 and oral etoposide on days 1-21 and 29-49 immediately followed by cisplatin IV over 1-2 hours on days 1-3 and 29-31. Treatment repeats every 8 weeks for 2 courses. Patients receive concurrent cranial radiotherapy daily over 8 weeks during course 2. Patients then receive carmustine IV over 1-2 hours every 8 weeks for 4 courses. Treatment continues in the absence of disease progression or unacceptable toxicity. Quality of life is assessed before the study, prior to each treatment course, every 4 months for 1 year, every 6 months for 4 years, and then annually for 5 years. Patients are followed every 4 months for 1 year, every 6 months for 4 years, annually for 5 years, and then for survival.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed newly diagnosed glioblastoma multiforme No oligodendrogliomas or oligoastrocytomas

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 130,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT no greater than 2 times ULN Renal: Creatinine no greater than 0.5 mg/dL above ULN Other: No uncontrolled infection No other major medical conditions No other concurrent malignancy except superficial skin cancers Must be able to read English (quality of life assessment only) No other problem that may preclude quality of life assessment Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Concurrent steroids allowed Radiotherapy: No prior radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 1999-05; Primary Completion 2001-08 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
overall survival | Up to 10 years

SECONDARY OUTCOMES:
quality of life | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J. Moynihan, MD, Study Chair — Mayo Clinic
Locations (19):
- United States (19):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Result] Jaeckle K, Ballman K, O'Fallon J, et al.: Response to pre-radiation chemotherapy as a predictor of survival in patients with newly diagnosed malignant astrocytoma: a North Central Cancer Treatment Group (NCCTG) study. [Abstract] Neuro-Oncology 6 (4): TA-26, 376, 2004.
- [Result] Jaeckle K, Ballman K, Uhm J, et al.: Relationship of administration of enzyme-inducing anticonvulsants (EIAC) to survival in patients with glioblastoma: a North Central Cancer Treatment Group (NCCTG) study. [Abstract] Neuro-Oncology 6 (4): TA-27, 376, 2004.